CLINICAL TRIAL: NCT04629053
Title: Determining the Causes and Outcomes of Febrile Illness in Health Care Facilities in Rural South and Southeast Asia, as Part of the South and Southeast Asian Community-based Trials Network (SEACTN). Work Package B (WP-B).
Brief Title: Causes and Outcomes of Febrile Illness in Health Facilities in Rural South and Southeast Asia
Acronym: SEACTN-WP-B
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Shoklo Malaria Research Unit (SMRU) (Unknown); Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other); Building Resources Across Communities (BRAC), Bangladesh (Unknown); Mahidol Oxford Tropical Medicine Research Unit (Other); Chiang Rai Clinical Research Unit (CCRU), Thailand (Unknown)
Responsible Party: Sponsor
Other Study IDs: BAC20003
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Febrile Illness
Keywords: Acute Febrile Illness; Causes; Outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples and nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an acute febrile illness: Patients with acute febrile illness, 4,800 children and 2,400 adults, divided equally across four countries (Laos, Myanmar,Thailand (including the Thai-Myanmar border region), and Bangladesh) and three age groups: >28 days to <5 years; ≥5 years to <15 years, and ≥15 years of age.

SUMMARY:
This prospective multi-site observational study aims to describe causes and clinical outcomes of acute febrile illness as well as host biomarkers in patients aged >28 days residing in rural areas in Laos, Myanmar, Thailand, the Thai-Myanmar border region, and Bangladesh and presenting with acute febrile illnesses (≤ 14 days duration) to participating health facilities.

This study is funded by the UK Wellcome Trust. The grant reference number is 215604/Z/19/Z

DETAILED DESCRIPTION:
The majority of people in low- and middle-income countries (LMICs) in South and Southeast Asia live in rural areas. These people are some of the poorest in the region and the exact health issues which concern them have not been well defined, in that they have not been fully studied. Despite this lack of data, there are indications that disease of an infectious aetiology, 'febrile illness,' in particular in the tropics, still accounts for significant morbidity and mortality. This is in contrast to higher-income countries.

The South and Southeast Asian Community-based Trials Network in Rural Febrile Illness project (SEACTN RFI) aims to better understand and quantify the burden of febrile illness, the aetiological causes and the manner in which it affects the people of the area, all on a scale which has not been attempted before. It will collect information to help better understand and predict these outcomes based on a multitude of factors, which will form the basis for interventions within the network in the future. The initial study will be observational, as the current understanding of the local health issues and the health systems in these areas is insufficient to know how best to intervene.

In a separate work package, Work Package A (WP-A), the investigators will be collecting data from within the participating SEACTN communities through village health workers (VHWs) and local health facilities on the incidence, causes and outcomes of febrile illness in these areas.

In Work Package B (WP-B) will recruit patients seeking care at higher level facilities than the WP-A VHWs and health centres. These patients are likely to be more severely ill, in order to obtain a more thorough understanding of the causes and burden of febrile illness in these areas. A broader range of specimens, including venous blood samples and respiratory specimens will be collected. In-depth diagnostic testing including blood cultures, serological assays, pathogen molecular diagnostics, host biomarker assays, and validation of pathogen-blind next generation sequencing approaches will be conducted. The data from WP-A gathered in the community complemented by the WP-B data from higher level health facilities in the same regions will provide a rich understanding of the causes, incidence and outcomes of febrile illness in these areas. These data will be analysed using advanced statistical methodology to create electronic decision-support tools (eDSTs) to aid VHWs in their assessment, triage and treatment of patients. These and other relevant interventions will later be trialled across the SEACTN villages.

ELIGIBILITY:
Inclusion Criteria:

1. The patient and/or where relevant their parent/guardian/caretaker is willing and able to give informed consent /assent for participation in the study;
2. Aged > 28 days (day of birth = Day 1);
3. Axillary temperature at presentation (≥ 37.5°C (99.5°F) OR < 35.5°C (95.9°F)) and no more likely cause than sepsis for hypothermia OR History of fever in the 24 hours prior to presentation;
4. Onset of illness ≤ 14 days

Exclusion Criteria:

1. Accident or trauma is the cause for the patient's presentation;
2. Presentation ≤ 3 days after routine immunisations
3. Is currently under follow-up or has been afebrile for less than 72 hours after completion of a follow-up period.
4. The treating healthcare worker's decision is to send the patient home following initial assessment.

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients residing in rural areas in Laos, Myanmar, Thailand, the Thai-Myanmar border region, and Bangladesh and presenting with acute febrile illnesses to participating health facilities
Sampling Method: Non-Probability Sample
Enrollment: 7200 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pathogens | Samples collected over approximately 1 month
  Prevalence of a range of pathogens identified from febrile patients, analysed by region and participant age group

SECONDARY OUTCOMES:
Recovery status | Approximately 1 month
  Recovery status e.g. full recovery, partial recovery, deterioration, and death at specified time points up to 28 days from enrolment
The association between host biomarkers and other predictors with aetiological diagnoses and clinical outcomes | Samples collected over approximately 1 month
  The area under the curve, sensitivity and specificity of host biomarkers and other predictors to identify bacterial infections and to predict severe outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Lubell, Prof., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (4):
- Building Resources Across Communities (BRAC), Dhaka, Bangladesh
- Laos-Oxford-Mahosot Wellcome Trust Research Unit, Vientiane, Laos
- Thailand (2):
  - Shoklo Malaria Research Unit, Mae Sot, Changwat Tak
  - Chiangrai Clinical Research Unit (CCRU), Chiang Rai

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)